CLINICAL TRIAL: NCT05894421
Title: Phase I Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of TQB2223 Injection Combined With Penpulimab Injection in Subjects With Advanced Cancers
Brief Title: TQB2223 Injection in Combination With Penpulimab in Patients With Advanced Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2223-I-01
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2223 injection+ Penpulimab Injection (Experimental): intravenous injection of TQB2223 injection and Penpulimab injection for one times every three weeks, 21 days as a treatment cycle.
  Interventions: Drug: TQB2223 injection+ Penpulimab Injection

INTERVENTIONS:
Drug: TQB2223 injection+ Penpulimab Injection — TQB2223 is an anti lymphocyte activation gene-3 (LAG-3) antibody. Penpulimab Injection is an anti-PD-1 antibody.

SUMMARY:
TQB2223 is a recombinant, fully humanized antibody that binds lymphocyte activation gene-3 (LAG-3) and blocks the LAG-3/ major histocompatibility complex class II (MHC-II) interaction, thus allowing for increased T-cell proliferation and cytokine production. This is a phase I study to evaluate the safety, tolerability, pharmacokinetics (PK) and effectiveness of TQB2223 injection in combination with Penpulimab in subjects with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Male or female patient 18 to 75 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥3 months;
* Histologically or cytologically confirmed malignancies;
* Subjects with advanced malignant tumors who failed standard treatment or lacked effective treatment;
* Patient has at least one evaluable lesion assessed by RECIST 1.1;
* The main organs function is well;
* Male or female patient had no plans to become pregnant and voluntarily take effective contraceptive measures during study period until at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Concurrent secondary malignancy. or other malignancy with no evidence of disease for more than 5 years;
* History of uncontrolled intercurrent illness;
* Major surgical procedure, radiotherapy, chemotherapy, or immunotherapy within 4 weeks prior to first dose;
* Prior treatment targeting LAG-3;
* Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first treatment cycle (21 days).
  DLT is defined as toxicities that meet pre-defined severity criteria of Common Terminology Criteria for Adverse Events (CTCAE) v5.0, and assessed as having a suspected relationship to TQB2223 injection, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (21 days) of treatment.
Maximum tolerated dose (MTD) | During the first treatment cycle (21 days).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks.
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria and Guidelines for Response Criteria for Use in Trials Testing Immunotherapeutics (iRECIST) for solid tumors, Lugano 2014 criteria and Lymphoma Response to Immunomodulatory therapy Criteria (LYRIC) for lymphoma.

SECONDARY OUTCOMES:
Percentage of anti-drug antibody (ADA) positive patients | Pre-dose on Cycle 1, 2, 4, 8 . 30 days and 90 days after the last dose. Each cycle is 21 days.
  Percentage of ADA positive patients will be calculated to evaluate immunogenicity of TQB2223.
The area under the curve (AUC) | 5 minutes, 2 hour, 6 hours, 24 hours, 144 hours and 336 hours after dose on cycle 1 and cycle 3. Pre-dose on cycle 2, 4, 5, 6, 7, 8. Each cycle is 21 days.
  The area under the curve (AUC) of serum concentration of TQB2223
Peak concentration (Cmax) | 5 minutes, 2 hour, 6 hours, 24 hours, 144 hours and 336 hours after dose on cycle 1 and cycle 3. Pre-dose on cycle 2, 4, 5, 6, 7, 8. Each cycle is 21 days.
  Maximum observed concentration (Cmax) of TQB2223
Terminal half-life (T1/2) | 5 minutes, 2 hour, 6 hours, 24 hours, 144 hours and 336 hours after dose on cycle 1 and cycle 3. Pre-dose on cycle 2, 4, 5, 6, 7, 8. Each cycle is 21 days.
  The terminal elimination half-life (t 1/2) is the time that takes for the elimination processes to reduce the plasma concentration of the drug in the body by 50 %.
Receptor occupation (RO) | 5 minutes, 2 hour, 6 hours, 24 hours, 144 hours and 336 hours after dose on cycle 1 and cycle 3. Pre-dose on cycle 2, 4, 5, 6, 7, 8. Each cycle is 21 days.
  Receptor occupation (RO) of LAG-3 after administration.
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria and Guidelines for Response Criteria for Use in Trials Testing Immunotherapeutics (iRECIST) for solid tumors, Lugano 2014 criteria and Lymphoma Response to Immunomodulatory therapy Criteria (LYRIC) for lymphoma.
Disease control rate (DCR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Defined as the proportion of subjects with CR, PR, or Stable Disease (SD).
Duration of Response (DOR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Defined as the time from first documented response to documented disease progression or death.
Progression-free survival (PFS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Defined as the time from the first dose of TQB2223 to the first occurrence of disease progression or death from any cause.
Overall survival (OS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Overall survival refers to the time from the first treatment to death from any cause.
Number of patients with adverse events (AEs) | From the time of informed consent signed to 28 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of patients with serious adverse events (SAEs) | From the time of informed consent signed to 28 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The second hospital of Dalian medical university, Dalian, Liaoning
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No